CLINICAL TRIAL: NCT03824210
Title: A Study to Co-produce, and Explore the Impact of, an App-based Support Intervention on Young Carers
Brief Title: A Study to Co-produce a Young Carers App
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RD2018-70
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Caring
MeSH Terms: interventions — Amyloid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stage 1: School children age 11-18 (from two nominated schools) and young carers 11-18
  Interventions: Other: App
- Stage 2: Young carers from Young Carers in Herts 11-18
  Interventions: Other: App

INTERVENTIONS:
Other: App — Mobile phone app

SUMMARY:
This study will co-produce and pilot-test a mobile phone App and a booklet, with input from local secondary schools and carer support groups to develop and pilot-test the App, in order to ensure it is designed to meet young people's needs. This App will serve to increase knowledge, information and provide strong links for young carers and local support available.This is a mixed methods study, using a transformative design. A transformative approach centres on users' needs and uses their experiences to shape how the App will look (in this case, uses are young carers). Carers will co-produce the App and booklet. The study will explore how a free app-based online support tool can help enhance support for young carers. Young carers have been involved since the outset and drove this planned study.

DETAILED DESCRIPTION:
This study will provide evidence about App usage in young carers (YCs), there is no evidence to date on this to the researcher's knowledge. While there are articles and reports on young carers and their experiences there is very little actual empirical research, partly due to the hard-to-reach population and their carer responsibilities and associated experiences (such as carer burden).

The study seeks to identify the gap between estimated and actual numbers of young carers, as part of Stage 3, which will again add to the evidence base as this has not previously been reported. The study will be able to describe the impact of a technology-based intervention to increase support for YCs.

This research will also contribute to understanding how App-based support can help YC, specifically exploring how receiving centralised, comprehensive information regarding: looking after their own health; having time off from carer duties and resources to support them getting this; self-awareness or self-identification of carer responsibilities and the impact of being a carer, might help.

Young Carers have also talked about the need for networks and support; these individuals will then be able to access Young Carers in Herts - and find support locally via professionals (they can access links to counsellors via the App -in order to receive mental health support) as well as other young carers (peer support, identified as very important in other recent local work).

This proposed research, through the qualitative interviews and focus groups, will also allow investigators to contribute an in-depth picture of (including a longitudinal description from the YCs in-depth interviews over the course of a year) of young carers' needs, and identify where needs are not being met and what could be done to improve their experiences. Having contextual data from interviews from peers (senior school age children), who may themselves end up becoming young carers, will also give us data to contrast.

This research will also help primary and secondary care providers to understand the needs and identification of this group. Although the study is not explicitly looking at this, the researchers hope to look at this in future work.

ELIGIBILITY:
Inclusion Criteria:

* School children from nominated schools in Hertfordshire (stage 1)
* Ability to provide informed consent (consent processes/literature will be age appropriate 11-17) (stage 2)
* Able to complete questionnaires (stage 2)

Exclusion Criteria:

* Does not speak or understand English
* Lacks mental capacity
* Young carers outside Hertfordshire

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young Carers in Hertfordshire
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
To understand young carer experiences, co-produce and develop an App for young carers 11yrs-18yrs age range in order to improve outcomes for family members and young carers | 18 months
  Measured by qualitative feedback on the app via transcriptions. Includes understanding of transition points such as admission/discharge to hospital.

SECONDARY OUTCOMES:
Formulation of a Young Carer Handbook | 18 months
  Co-creation of a Young Carer Handbook
Gain understanding of App usage | 18 months
  Number of views and downloads
Explore usefulness of the App and experience of caring over time | 18 months
  Transcripts of qualitative feedback
Capture information on referral rates of Young Carers before and after App introduction | 18 months
  Number of referrals of Young carers in Herts

CONTACTS AND LOCATIONS:
Locations (1):
- East and North Hertfordshire NHS Trust, Stevenage, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Identifiable data will not be shared with other researchers. The publication plan in the study protocol will be followed.